CLINICAL TRIAL: NCT05102851
Title: Impact of Prediabetes On Acute Coronary Syndrome in Sohag University Hospital
Brief Title: Impact of Prediabetes on Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Dina Abdelnasser Elamir, Resident doctor at Internal Medicine department, Sohag University Hospital, Sohag University
Other Study IDs: Soh-Med-21-07-05
Record Dates: First submitted 2021-08-18; First posted 2021-11-02 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2021-07

CONDITIONS: Diabetic Cardiomyopathy
MeSH Terms: conditions — Diabetic Cardiomyopathies | interventions — Body Mass Index

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with acute coronary syndrome: All patients with the acute coronary syndrome were included in the study. Pre-diabetic patient. Non-diabetic patient(Controlled)
  Interventions: Diagnostic Test: Troponin, Lipid profile, HBA1C, Fasting blood glucose level, Creatinine, Body Mass Index

INTERVENTIONS:
Diagnostic Test: Troponin, Lipid profile, HBA1C, Fasting blood glucose level, Creatinine, Body Mass Index — Full history: age, sex, smoking, known diabetes, positive family history high serum creatinine, history of prior percutaneous coronary intervention (PCI) or coronary arteries bypass grafting (CABG), or acute coronary syndrome (ACS). hypertension, diet.

SUMMARY:
Diabetes mellitus is one of the chronic non-communicable diseases which have emerged as a leading global health problem. According to the International Diabetes Federation Atlas guideline report, currently, there are 352 million adults with impaired glucose tolerance who are at high risk of developing diabetes in the future. In 2017, it was estimated that 425 million people (20-79 years of age) suffered from Diabetes mellitus, and the number is expected to rise to 629 million by 2045. Moreover, Egypt is considered one of the top 10 countries in the world

DETAILED DESCRIPTION:
Acute Coronary Syndrome refers to a constellation of symptoms compatible with acute myocardial ischemia. The syndrome includes systolic time segment elevation myocardial infarction non-systolic time segment elevation myocardial infarction and unstable angina.

Patients have an over tenfold risk for cardiovascular disease in their lifetime. In the United States, 77% of diabetes-related hospital admissions are for cardiovascular complications. A key feature of diabetes contributing to this is the development of accelerated atherosclerosis.

Prediabetes is a collective term that encloses individuals with glucose levels lower than cutoff levels for diabetes but too high to be considered normal. Fasting blood glucose 6.1 mmol/L- <7.0 mmol/L. In impaired glucose tolerance the ranges of blood glucose are>7.8 mmol/L-<11.1 mmol/L4.

Prediabetes is associated with a significant increase in cardiovascular morbidity and mortality and necessitates early and adequate intervention to prevent the development of complications, and progression to overt diabetes.

Higher fasting glucose levels in patients with the acute coronary syndrome were associated with worse clinical outcomes irrespective of the presence of diabetes mellitus. Similarly, higher fasting glucose was a marker of adverse outcomes in patients without diabetes presenting with acute systolic time segment elevation myocardial infarction.

Impaired glucose tolerance is common among non-diabetic patients admitted with the acute coronary syndrome. However, evidence is controversial regarding the prognostic impact of 'prediabetes' on the clinical outcome

ELIGIBILITY:
Inclusion Criteria:

* All patients with acute coronary syndrome
* Diabetic patients and will be subdivided into controlled and uncontrolled Pre-diabetic patients.
* Non-diabetic patient(Controlled)

Exclusion Criteria:

* Patient under 18 years old
* Pregnancy
* Chronic kidney disease
* Familiar hyperlipidemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Statistical presentation and analysis of the present study will be conducted SPSS V.22. Data will be expressed into phases:
  Ι- Descriptive Mean value(X) and Standard Deviation (SD): for quantitative data. Frequency and percentage for qualitative data.
  Π- Analytic by t-student test and Chi-square test. P value >0.05 will be considered statistically non-significant. P value ≤0.05 will be considered statistically significant.
  P value ≤0.001 will be considered statistically highly significant. Variance: Correlation of MPV with other parameters was performed by Pearson correlation test (r value as the coefficient).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Hba1c | Day 1
  We consider patients with Hba1c less than 5.7% not diabetic , Patients with Hba1c from 5.7%-6.4% prediabetic and patients with Hba1c 6.5% or more diabetic patients
CCU admission | 6 months
  All patients admitted with acute coronary syndrome will be included in the research

CONTACTS AND LOCATIONS:
Overall Officials: Amal K. Ahmed, Ass. Prof., Study Director — Sohag University; Hany A. Muhammed Khalil, Lecturer, Study Chair — Sohag University
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided